CLINICAL TRIAL: NCT03057353
Title: Risk Factors for Ligamentum Flavum Hypertrophy in Lumbar Spinal Stenosis Patients From Xinjiang Uygur Autonomous Region of China: a Retrospective, Single-center, Case Analysis
Brief Title: Risk Factors for Ligamentum Flavum Hypertrophy in Lumbar Spinal Stenosis Patients
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Sixth Affiliated Hospital of Xinjiang Medical University (Other)
Responsible Party: Principal Investigator, Gang Zhou, Attending Physician, Sixth Affiliated Hospital of Xinjiang Medical University
Other Study IDs: SixthAHXinjiang_01
Record Dates: First submitted 2017-02-15; First posted 2017-02-20 (Actual); Last update posted 2017-02-20 (Actual); Status verified 2017-02

CONDITIONS: Lumbar Spinal Stenosis
MeSH Terms: conditions — Spinal Stenosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- lumbar CT imaging: Collecting lumbar CT imaging data of 104 patients with lumbar spinal stenosis to observed the incidence of ligamentum flavum hypertrophy of patients with different nationalities, sexes, heights, ages, and weights and explored risk factors affecting ligamentum flavum hypertrophy.
  Interventions: Device: lumbar CT imaging

INTERVENTIONS:
Device: lumbar CT imaging — Collecting lumbar CT imaging data of 104 patients with lumbar spinal stenosis to observed the incidence of ligamentum flavum hypertrophy of patients with different nationalities, sexes, heights, ages, and weights and explored risk factors affecting ligamentum flavum hypertrophy.

SUMMARY:
To measure ligamentum flavum thickness in patients with different nationalities, sexes, heights, ages, and weights from Xinjiang Uygur Autonomous Region of China with CT, explore the correlation between various factors and ligamentum flavum thickness, provide reference for pedicle screw placement and lumbar decompression surgery, develop individualized surgical programs, and can effectively reduce the incidence of unnecessary postoperative complications induced by misplacement.

DETAILED DESCRIPTION:
History and current related studies With the increase of human social activities, spinal degenerative disease is increasing year by year. Due to the special anatomical structures and biomechanical characteristics, lumbar vertebrae easily suffer from lumbar spinal stenosis. Lumbar spinal stenosis is a medical condition in which the spinal canal narrows and compresses the spinal cord and nerves at the level of the lumbar vertebra. Vertebral spondylolisthesis, facet joint hyperplasia, bony spur posterior extension, intervertebral disc prolapse/protrusion, and ligamentum flavum hypertrophy are common causes for degenerative lumbar spinal stenosis, and ligamentum flavum hypertrophy is one of the important causes for spinal stenosis. When conservative treatment is ineffective, the occurrence of muscle paralysis or bladder symptoms caused by nerve compression requires surgical treatment. Commonly used surgical methods include pedicle screw fixation, flavectomy, laminectomy and facetectomy. Therefore, important anatomical structures will be involved in the operation, such as pedicle, ligamentum flavum, lamina, and articular process.

Many previous studies concern pedicle morphology, lumbar ligamentum flavum, lamina and articular process, and important reference data are listed in Table 1. Safak et al. verified that ligamenta flavum thickness was not associated with sex; ligamenta flavum was remarkably thicker on the left side of segments L4/5 and L5/S1 than that on the right side; ligamenta flavum thickness was not positively correlated with age. Few studies address whether ligamenta flavum thickness was associated with nationality, sex and obesity.

Data collection, management, analysis and open-access

1. Written and electronic data were collected. The electronic data were stored in a specialized computer, and locked by the data manager. The written data were stored and locked in a reference room. The key was kept by the data manager and laboratory manager.
2. The locked database was not altered and was preserved, along with the original records. The database was statistically analyzed by a professional statistician.
3. Prior to any analysis of the data, the analysis plan outlined in this section would be reviewed, and detailed statistical analysis plans would be prepared and approved. All data regarding this trial were preserved by the Sixth Affiliated Hospital, Xinjiang Medical University, China.
4. Anonymized trial data would be published at www.figshare.com.

Statistical analysis

1. All data were analyzed using SPSS 21.0 software (IBM, Armonk, NY, USA).
2. All measurement data were normally distributed and expressed as mean ± standard deviation.
3. Ligamentum flavum thickness was compared among groups using two-sample t-test or one-way analysis of variance. Paired comparison between groups was conducted using Student-Newman-Keuls test. Correlation of nationality, sex, height, age and weight with ligamentum flavum thickness was analyzed using Pearson's correlation coefficient. Risk factors for ligamentum flavum hypertrophy were analyzed using multiple linear regression analysis. Odd ratio and 95% confidence interval were calculated.
4. The significance level was α = 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Lumbar spinal stenosis revealed by Lumbar CT images
* Complained of low back pain
* Age between 45 and 80 years old
* Irrespective of sex
* Signed informed consent

Exclusion Criteria:

* Spinal injury
* Spinal tumor
* Spinal infection
* Congenital or acquired spine deformity
* Pulmonary tuberculosis
* Severe systemic disease such as malignant tumor
* Cannot cope with the doctor due to mental illness or other causes

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 104 patients were evaluated after they signed the informed consent, including sex, age, height, nationality, weight, history of present illness, past history, family history, personal history, marital history, laboratory examination, and CT examination.
Sampling Method: Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2012-05 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Ligamentum flavum thickness | from May 2012 to May 2016
  Changes in ligamentum flavum thickness were observed under different influential factors.

SECONDARY OUTCOMES:
Lumbar morphology of patients | from May 2012 to May 2016
  Changes in ligamentum flavum morphology.

CONTACTS AND LOCATIONS:
Overall Officials: Gang Zhou, Master, Principal Investigator — Sixth Affiliated Hospital of Xinjiang Medical University

IPD SHARING:
Plan to Share IPD: Undecided